CLINICAL TRIAL: NCT07391098
Title: Peripheral Perfusion and Outcomes in ICU Patients With Sepsis (PERFUSE-ICU)
Brief Title: Peripheral Perfusion and Outcomes in ICU Patients With Sepsis
Acronym: PERFUSE-ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Alexandra Elena Lazăr (Other)
Responsible Party: Sponsor-Investigator, Alexandra Elena Lazăr, Associate prof, George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures
Organization: George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other)
Other Study IDs: GEPaladeU
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: SEPSIS; Septic Patients
Keywords: Peripheral perfusion; Capillary refill time; Veno-arterial carbon dioxide difference; Sepsis outcomes; Tissue hypoperfusion; Intensive care unit; Veno-arterial carbon dioxide difference ΔCO₂ gap
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SEPTIC PATIENTS: This cohort includes adult participants admitted to the intensive care unit with sepsis or septic shock, defined according to Sepsis-3 criteria with a Sequential Organ Failure Assessment (SOFA) score of 2 or higher at inclusion.
  Participants will receive standard ICU care according to local protocols. Peripheral perfusion will be assessed using capillary refill time and end-tidal carbon dioxide measurements at predefined time points (baseline, 6 hours, and 24 hours). In addition, paired arterial and venous blood gas samples will be collected at the same time points to evaluate markers of tissue perfusion, including lactate levels and the veno-arterial carbon dioxide difference.
  No experimental treatments or protocol-driven changes to clinical management will be introduced.
  Interventions: Other: PERIPHERAL PERFUSION EVALUATION

INTERVENTIONS:
Other: PERIPHERAL PERFUSION EVALUATION — This intervention consists of a predefined, multimodal peripheral perfusion assessment combining bedside clinical evaluation and blood gas analysis. Capillary refill time is measured at standardized time points, together with concurrent end-tidal carbon dioxide recording. Paired arterial and venous blood gas samples are obtained at the same time points to calculate the veno-arterial carbon dioxide difference and assess lactate levels. The intervention is limited to repeated physiological measurements during the first 24 hours of ICU admission and does not include any therapeutic intervention or protocol-driven change in clinical management

SUMMARY:
People with sepsis who are treated in the intensive care unit (ICU) often have impaired blood flow to the skin and other tissues. These alterations in tissue perfusion may be associated with disease severity and clinical outcomes.

The aim of this study is to see whether simple signs of blood flow to the skin, such as capillary refill time and blood test measurements, are linked to outcomes in people with sepsis treated in the ICU.

Adults with sepsis who are admitted to the ICU will be invited to take part. Researchers will collect routine clinical data and blood test results during the first day of ICU treatment. No extra procedures or treatments will be performed as part of the study.

The results of this study may improve understanding of early signs of impaired circulation in sepsis and their relation with recovery and survival.

DETAILED DESCRIPTION:
Sepsis is a life-threatening condition caused by a dysregulated host response to infection and is associated with high morbidity and mortality in intensive care units (ICUs). Early detection of impaired tissue perfusion is essential for risk stratification and may help predict clinical outcomes.

Peripheral perfusion can be assessed using a combination of bedside clinical signs and physiological and biochemical markers. Capillary refill time (CRT) is a simple, non-invasive bedside measure of peripheral perfusion. In addition, respiratory and blood gas-derived variables, such as end-tidal carbon dioxide (ETCO₂) and the veno-arterial carbon dioxide difference (ΔCO₂), may reflect alterations in tissue blood flow and microcirculatory dysfunction. However, the relationship between these markers and clinical outcomes in patients with sepsis is not fully established.

This is a prospective observational cohort study conducted in adult ICU patients with sepsis or septic shock. Eligible participants will be enrolled after ICU admission. Sepsis will be defined according to Sepsis-3 criteria, with a Sequential Organ Failure Assessment (SOFA) score of 2 or higher at inclusion. Baseline disease severity will be further assessed using the Acute Physiology And Chronic Health Evaluation (APACHE) IV score.

Peripheral perfusion markers will be recorded at predefined time points: at inclusion (T0), six hours (T6), and twenty-four hours (T24). CRT and ETCO₂ will be measured at the bedside, using standardized methods. Arterial and venous blood gas samples will be obtained at the same time points to determine PaCO₂, PvCO₂, lactate levels, and the veno-arterial carbon dioxide difference (ΔCO₂). Blood sampling will be performed through existing arterial or venous catheters whenever possible.

Additional routinely collected clinical data will include hemodynamic variables, ventilatory parameters, vasopressor use, and organ support. Outcomes will include SOFA score on day three, ventilator-free days and vasopressor-free days within the first seven days, and vital status at day 7 and day 28.

No experimental treatments or protocol-driven changes to standard clinical management will be introduced. This study aims to evaluate the association between early peripheral perfusion markers-combining CRT, ETCO₂, and blood gas-derived variables-and short-term outcomes in adults with sepsis treated in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years or older
* admission to the intensive care unit
* sepsis or septic shock, defined according to Sepsis-3 criteria
* SOFA score ≥ 2 at inclusion
* presence of an arterial line and a central venous catheter suitable for blood sampling
* possibility to perform peripheral perfusion assessment (CRT) at predefined time points

Exclusion Criteria:

* age under 18 years
* pregnancy
* expected ICU stay less than 24 hours
* limitations of therapy at ICU admission (e.g., DNR or comfort-only care)
* improper central venous catheter position (catheter tip not located in the superior vena cava)
* absence of arterial or central venous access required for paired blood gas sampling
* refusal of consent, when applicable according to local ethics requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult patients admitted to the intensive care unit with sepsis or septic shock, defined according to Sepsis-3 criteria, with a Sequential Organ Failure Assessment (SOFA) score of ≥ 2 at the time of inclusion. Participants will be enrolled early after ICU admission and managed according to standard care and local treatment protocols.
  The study population consists of critically ill patients requiring invasive monitoring, enabling the assessment of peripheral perfusion using capillary refill time and paired arterial and venous blood gas analyses during the first 24 hours of ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Sequential Organ Failure Assessment (SOFA) score from inclusion (day 0) to day 3. | From enrollemnt to day 3
  The SOFA score ranges from 0 to 24, with higher scores indicating greater organ dysfunction and worse clinical status.
  The change score is calculated as SOFA score at day 3 minus SOFA score at inclusion, with positive values indicating worsening organ dysfunction and negative values indicating improvement.

SECONDARY OUTCOMES:
Ventilator-Free Days (0-7) | first 7 days
  Ventilator-free survival days from day 0 to day 7, with death before day 7 assigned a value of 0.
Vasopressor-Free Days (0-7) | first 7 days
  Vasopressor-free survival days from day 0 to day 7 (death before day 7 scored as 0).
Vital Status on Day 7 | first 7 days
  Survivor or non-survivor at day 7 after ICU admission.
Vital Status on Day 28 | first 28 days
  Survivor or non-survivor at day 28 after ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Elena Lazăr, Principal Investigator — George Emil Palade University of Medicine, Pharmacy, Science and Technology from Tirgu Mures, Romania
Locations (1):
- Emergebcy Clinical County Hospital - Intensive Care Clinic, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Undecided